CLINICAL TRIAL: NCT06322017
Title: Prospective Multicenter Randomized and Controlled Study Evaluating the Benefit of Early Pulmonary Vein Isolation Compared to Usual Treatment in Patients Aged Over 75 Years and Presenting With Atrial Fibrillation
Acronym: EDearly AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0450
Record Dates: First submitted 2024-02-08; First posted 2024-03-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Pulmonary vein isolation; Elderly Conventional management; Frailty
MeSH Terms: conditions — Atrial Fibrillation; Frailty | interventions — Flecainide; Sotalol; Amiodarone; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rhythm control by Pulmonary Vein Isolation (PVI) procedure (Experimental)
  Interventions: Procedure: Rhythm control by Pulmonary Vein Isolation (PVI) procedure
- Conventional care by antiarrhythmic drugs or bradycardic drugs (Active Comparator)
  Interventions: Drug: Conventional care by antiarrhythmic drugs (flecainide, sotalol, amiodarone) or bradycardic drugs (all betablocker or calcium channel blocker therapy, digoxin)

INTERVENTIONS:
Procedure: Rhythm control by Pulmonary Vein Isolation (PVI) procedure — The PVI procedure involves the creation of a circumferential lesion around the ostium of the four pulmonary veins.
  The choice of the type of energy to insure the lesion will be left to the discretion of the investigator, according to the center's habits and the patient's anatomy found on the scanner.
  Arms: Rhythm control by Pulmonary Vein Isolation (PVI) procedure
Drug: Conventional care by antiarrhythmic drugs (flecainide, sotalol, amiodarone) or bradycardic drugs (all betablocker or calcium channel blocker therapy, digoxin) — Ventricular rate control is carried out using negative chronotropic agents (e.g. beta-blockers, calcium channel blockers, digitalis, etc.) according to current recommendations. If this fails, ablation of the atrioventricular junction with placement of a permanent pacemaker can be carried out according to current recommendations. As part of this research, the choice of bradycardic drugs and interventions will be left to the discretion of the investigator according to the center's practices and current recommendations.
  Rhythm control aims to reduce AF by cardioversion (if it persists) to restore sinus rhythm and subsequently maintain it by introducing anti-arrhythmic treatment. Several antiarrhythmic drugs (flecainide, sotalol or amiodarone) can be used in this setting. As part of this research, the choice of antiarrhythmic drugs will be left to the discretion of the investigator according to the center's practices and current recommendations.
  Arms: Conventional care by antiarrhythmic drugs or bradycardic drugs

SUMMARY:
Therapeutic management of Atrial Fibrillation (AF) is based either on heart rate control or on rhythm control, a strategy which aims to maintain a normal heart rhythm. The benefit in terms of morbidity and mortality of a normal heart rhythm would, however, be largely offset by the frequent side effects of antiarrhythmic drugs which could even lead to an increase in mortality compared to rate control. This increase has particularly been suggested in people aged over 75.

Since the emergence of catheter Pulmonary Vein Isolation (PVI), an effective alternative to antiarrhythmic drugs has become available. This technique makes it possible to isolate the foci triggering AF under local or general anesthesia with greater effectiveness than medications and very low risks. Records in the elderly do not seem to show a reduction in effectiveness or an increase in complications. However, in the absence of a dedicated randomized study, its use is strongly limited in the elderly where rate control (52% of people over 65 years old) and the use of antiarrhythmic drugs are largely favored due to the simplicity of implementation and the low cost of medications.

However, an early rhythm control strategy seems to reduce cardiovascular events in relatively old individuals (average age 70 years). The use of PVI in first line could make it possible to further improve these results.

The objective of the investigator is therefore to carry out the first randomized comparative study proposing to evaluate the impact of early PVI compared to usual treatment in patients aged 75 and over with AF.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 75 and over.
* Paroxysmal AF or early recurrent or persistent paroxysmal AF first diagnosed less than 12 months ago.
* Patient who consented to participate in the study.
* Patient affiliated to a social security system.

Exclusion Criteria:

* Indication of cardiac pacing or defibrillation at baseline.
* History of valve replacement, atrial occlusion or exclusion.
* History of AF ablation.
* Contraindication to anticoagulation or an invasive procedure.
* Significant heart disease (structural with alteration of LVEF <35%, congenital heart disease, hypertrophic heart disease with wall of more than 15 mm, revascularized coronary syndrome less than 3 months old).
* Stroke less than 6 months old.
* Uncontrolled dysthyroidism.
* Chronic renal failure (CKD - eGFR <30 µMol/L).
* Patient under curatorship, guardianship, safeguard of justice.
* Life expectancy less than 24 months.
* Participation in another therapeutic trial likely to impact the study evaluation criteria.
* Severe cognitive impairment noted in history.
* Lack of understanding of the study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2030-04-09 (Estimated); Study Completion 2030-04-09 (Estimated)

PRIMARY OUTCOMES:
Time before occurrence of the first event among cardiovascular death, hospitalization (all causes) and stroke | 2 years
  Days

SECONDARY OUTCOMES:
Number of PVI peri-procedural complications | 48 hours
Number of complications | 2 years
Quality of life score | Inclusion
  EQ-5D-5L score
Quality of life score | 3 months
  EQ-5D-5L score
Quality of life score | 6 months
  EQ-5D-5L score
Quality of life score | 12 months
  EQ-5D-5L score
Quality of life score | 18 months
  EQ-5D-5L score
Quality of life score | 24 months
  EQ-5D-5L score
Number of documented episodes of AF | 2 years
Number of patients treated by cardiovascular drugs | 2 years
Doses of cardiovascular drugs | 2 years
  milligrams
Autonomy score | Inclusion
  Activities of Daily Living (ADL) score
Autonomy score | 3 months
  ADL score
Autonomy score | 6 months
  ADL score
Autonomy score | 12 months
  ADL score
Autonomy score | 18 months
  ADL score
Autonomy score | 24 months
  ADL score
Autonomy score | Inclusion
  Instrumental Activities of Daily Living (IADL) score
Autonomy score | 3 months
  IADL score
Autonomy score | 6 months
  IADL score
Autonomy score | 12 months
  IADL score
Autonomy score | 18 months
  IADL score
Autonomy score | 24 months
  IADL score
Body weight | Inclusion
  kilograms
Body weight | 3 months
  kilograms
Body weight | 6 months
  kilograms
Body weight | 12 months
  kilograms
Body weight | 18 months
  kilograms
Body weight | 24 months
  kilograms
Numbers of falls | Inclusion
Numbers of falls | 3 months
Numbers of falls | 6 months
Numbers of falls | 12 months
Numbers of falls | 18 months
Numbers of falls | 24 months
Physical performance score | Inclusion
  Short Physical Performance Battery (SPPB) test score
Physical performance score | 2 years
  SPPB test score
Evolution of ADL score according to the results of the Integrated Care for Older People (ICOPE) test at inclusion | 2 years
Evolution of IADL score according to the results of the ICOPE test at inclusion | 2 years
Cognitive assessment | Inclusion
  Mini-Mental State Examination (MMSE) score
Cognitive assessment | 2 years
  MMSE score
Cognitive assessment | Inclusion
  Batterie Rapide d'Efficience Frontale (BREF) score
Cognitive assessment | 2 years
  BREF score
Cognitive assessment | Inclusion
  Mini Geriatric Depression Scale (GDS) score
Cognitive assessment | 2 years
  Mini GDS score

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Gourraud, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire Atlantique, France

IPD SHARING:
Plan to Share IPD: No